CLINICAL TRIAL: NCT02643641
Title: Study to Evaluate the Effect of Different Pre-seasonal BM32 Dosing Schedules on the Rapid Induction of a Protective IgG Immune Response
Brief Title: Effect of Different Pre-seasonal BM32 Dosings on the Induction of a Protective Immune Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biomay AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CS-BM32-004
Record Dates: First submitted 2015-12-17; First posted 2015-12-31 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Hypersensitivity
Keywords: Grass pollen allergy; subcutaneous immunotherapy; allergy vaccine; dose regimen
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- BM32-3 (Experimental): 2 placebo injections will be given followed by 3 injections with 20 micrograms each of BM321, BM322, BM325 and BM326
  Interventions: Biological: BM32
- BM32-4 (Experimental): 1 placebo injections will be given followed by 4 injections with 20 micrograms each of BM321, BM322, BM325 and BM326
  Interventions: Biological: BM32
- BM32-5 (Experimental): 5 injections with 20 micrograms each of BM321, BM322, BM325 and BM326 will be given
  Interventions: Biological: BM32
- Placebo (Placebo Comparator): 5 placebo injections (alhydrogel only) will be given
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: BM32 — BM32 is a mixture of 4 different recombinant proteins directed at the major grass pollen allergens, adsorbed on aluminum hydroxide
  Arms: BM32-3; BM32-4; BM32-5
Biological: Placebo — Placebo contains aluminum hydroxide only
  Arms: Placebo

SUMMARY:
BM32 is a product for immunotherapy of grass pollen allergies. It consists of 4 different recombinant proteins (BM321, BM322, BM325 and BM326) adsorbed on alhydrogel. This prospective, double-blind. placebo controlled, mono-centric trial investigates the levels of allergen specific IgG antibodies following 3, 4 or 5 subcutaneous injections before the grass pollen season.

DETAILED DESCRIPTION:
The aim of this study is to further optimize the immunization schedule by

* moving the last injection into beginning of the grass pollen season for all study arms in order to ensure highest possible IgG4 levels when they are needed - i.e. at the peak of the grass pollen season,
* administration of more than 3 pre-seasonal injections in order to build up sufficiently high levels of IgG4 already in the first year of treatment , and
* dosing during the beginning of the grass pollen season to establish safety in this setting The effect of such optimized immunization schedule on the induction of an IgG4 immune response as a surrogate parameter for efficacy will be studied. The Total Nasal Symptom Score (TNSS) before and after the treatment and Combined Symptom-Medication Score (SMS) during the grass pollen season will be evaluated as secondary endpoints. This will allow intra-individual comparison of seasonal symptom data and responsiveness in the chamber setting.

ELIGIBILITY:
Inclusion Criteria:

* The subjects are grass pollen allergic but otherwise healthy. Healthy subjects are defined as individuals who are free from clinically significant illness or disease as determined by their medical history (including family), physical examination, laboratory studies, and other tests.
* They are aged 18 to 60 years inclusive.
* They have a history of seasonal allergic rhinitis (SAR) to grass pollen.
* They have a normal electrocardiogram without clinically significant abnormalities.
* They exhibit a moderate to severe response to approximately 1500 grass pollen grains/m3 after the first 2h in the Vienna Challenge Chamber, which is defined as a nasal symptom score (TNSS) of at least 6. (Nasal symptom score is the sum of nasal obstruction, rhinorrhoea, itchy nose and sneezing, each of which have been scored on a scale from 0 to 3).
* They have a positive skin prick test with a wheal diameter >5mm for grass pollen extract at the screening visit.
* They have a positive serum IgE test for timothy grass pollen and to rPhl p 1+rPhl p 5 at the screening visit (ImmunoCAP ≥3.5 kUA/l; i.e ≥ class 2)..
* There are no conditions or factors which would make the subject unlikely to be able to stay in the chamber for 6 hours.
* They are capable of giving informed consent which includes compliance with the requirements and restrictions listed in the consent form.
* They are available to complete all study measurements

Exclusion Criteria:

* Sensitization to Phl p 7
* Pregnant, lactating or sexually active women with childbearing potential who are not using a medically accepted birth control method (pregnancy to be controlled by a pregnancy dipstick test).
* On examination the subject is found to have any structural nasal abnormalities or nasal polyposis, a history of frequent nosebleeds, recent nasal surgery or ongoing upper respiratory tract infection which in the Responsible Physician's opinion renders the subject unsuitable for participation in the study.
* Any respiratory disease other than mild stable asthma that is controlled with occasional use of as-needed short-acting beta-agonists and associated with normal lung function.
* The subject is concurrently participating or has participated in any clinical study in the previous month.
* Participation in a SIT trial for grass pollen allergy in the three years prior to this study.
* Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease, endocrine disease or pulmonary disease (including but not confined to chronic bronchitis, emphysema, bronchiectasis or pulmonary fibrosis).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Titer of allergen specific IgG4 antibodies | approximately 6 months

SECONDARY OUTCOMES:
Total nasal symptom score upon pollen challenge (TNSS) | Change from baseline at 9 months
  Sensitivity to a grass pollen challenge in an environmental exposure chamber
Mean daily combined symptom and medication score (SMS) | 2 weeks
Well-being via visual analog scale | 2 weeks
Titers of allergen specific IgG antibodies | Up to 9 months

OTHER OUTCOMES:
Incidence of treatment emerging adverse events | up to 9 months
  Frequency and severity of IMP related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Petra Zieglmayer, MD, Principal Investigator — Vienna Challenge Chamber GmbH
Locations (1):
- Vienna Challenge Chamber, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes